CLINICAL TRIAL: NCT04500392
Title: High-flow Nasal Cannula Oxygenation Decrease Hypoxia in Sedated Gastrointestinal Endoscopes in Obesity: a Randomized Multicenter Clinical Trial
Brief Title: High-flow Nasal Cannula Oxygenation Decrease Hypoxia in Sedated Gastrointestinal Endoscopes in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai Oriental Hospital, Tongji University School of Medicine (Unknown)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HFNOIO
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hypoxia; Gastric Cancer; Esophagus Cancer; Polyp of Colon; Colon Cancer
Keywords: Hypoxia; Gastrointestinal endoscopes; High-flow nasal cannula Oxygenation
MeSH Terms: conditions — Hypoxia; Stomach Neoplasms; Esophageal Neoplasms; Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Oxygen(up to 6L/min) supplied with a regular nasal catheter
  Interventions: Device: Regular nasal cannula
- High-flow nasal cannula group (Experimental): Oxygen(up to 60L/min) supplied with high-flow nasal cannula
  Interventions: Device: High-flow nasal cannula oxygenation

INTERVENTIONS:
Device: High-flow nasal cannula oxygenation — Oxygen is supplied with a high-flow nasal cannula oxygenation device#the flow is up to 60L/min
  Arms: High-flow nasal cannula group
Device: Regular nasal cannula — Oxygen is supplied with a regular nasal cannula #the flow is up to 6L/min
  Arms: Control group

SUMMARY:
Hypoxia is the most common adverse event during gastrointestinal endoscopes sedated with propofol and sufentanil, especially in obese people. In the present study, high-flow nasal cannula oxygenation will be utilized in order to reduce the incidence of hypoxia among obesity.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing gastrointestinal endoscopes
* age≥18 years old and ≤70 years old
* patients or family members signed informed consent form
* ASA classification I-II
* BMI≥ 28kg/m²

Exclusion Criteria:

* Coagulation disorders or a tendency of nose bleeding;
* An episode/exacerbation of congestive heart failure (CHF) that requires a change in medication, diet or hospitalization from any cause in the last 6 months;
* Severe aortic stenosis or mitral stenosis;
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months;
* Acute myocardial infarction in the last 6 months;
* Acute arrhythmia (including any tachycardia - or bradycardia) with the fluid of hemodynamics instability;
* Diagnosed chronic obstructive pulmonary disease or current other acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy);
* Increased intracranial pressure;
* ASA classification Ⅲ-Ⅳ ;
* Mouth, nose, or throat infection;
* Liver and kidney disease
* Fever, defined as core body temperature > 37.5℃;
* Pregnancy, breastfeeding or positive pregnancy test;
* Emergency procedure;
* Patients or family members refused to participate
* Mental disorders and people without civil capacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours]
  (75% ≤ SpO2 < 90% for <60 s)

SECONDARY OUTCOMES:
The incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (90% ≤ SpO2 < 95%)
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  (SpO2 < 75% for any duration or 75% < SpO2 < 90% for >/=60 s)
Other adverse events include other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force and HFNC supportive oxygen therapy-related adverse events. | Patients will be followed for the duration of hospital stay, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Principal Investigator — Renji Hospital, Shanghai Jiaotong University, Shanghai, China
Locations (3):
- China (3):
  - Shanghai Tongji Hospital, Shanghai, Shanghai, China
  - Shanghai Oriental Hospital, Shanghai, Shanghai, China
  - Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai, China

REFERENCES:
- [Derived] Wang L, Zhang Y, Han D, Wei M, Zhang J, Cheng X, Zhang Y, Shi M, Song Z, Wang X, Zhang X, Su D. Effect of high flow nasal cannula oxygenation on incidence of hypoxia during sedated gastrointestinal endoscopy in patients with obesity: multicentre randomised controlled trial. BMJ. 2025 Feb 11;388:e080795. doi: 10.1136/bmj-2024-080795. PMID 39933757